CLINICAL TRIAL: NCT02598674
Title: Long Term Impact of Pediatric Acute Renal Injury in Severe Sepsis in in Children - IMPRESS-C
Brief Title: Severe Sepsis in Children - IMPRESS-C
Acronym: IMPRESS-C
Status: Withdrawn | Type: Observational
Why Stopped: Expired IRB
Sponsor: University of Florida (Other)
Collaborators: American Society of Nephrology (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500264
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease; Hypertension
Keywords: acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Hypertension | interventions — Iodohippuric Acid; Gadolinium; Glomerular Filtration Rate; Filtration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis with Severe AKI: This group will have a history of pediatric admission with sepsis-related Acute Kidney Injury (sAKI) which lead to classification of "injury" or "failure". The following test will be performed: urinary and serum studies to measure glomerular filtration rate by using gadolinium, renal plasma flow by using an injection of non-radioactive iodohippurate, followed by cardiovascular assessments using 24 hour ambulatory blood pressure monitoring, peripheral arterial tonometry and pulse wave velocities (PWV).
  Interventions: Drug: Iodohippurate; Procedure: 24 hour ambulatory Blood Pressure; Procedure: Peripheral Arterial Tonometry; Procedure: Pulse Wave Velocity; Drug: Gadolinium
- Control: This group will not have a history of pediatric admission with sepsis-related Acute Kidney Injury (sAKI). The following test will be performed: urinary and serum studies to measure glomerular filtration rate by using gadolinium, followed by cardiovascular assessments using 24 hour ambulatory blood pressure monitoring, peripheral arterial tonometry and pulse wave velocities (PWV).
  Interventions: Procedure: 24 hour ambulatory Blood Pressure; Procedure: Peripheral Arterial Tonometry; Procedure: Pulse Wave Velocity; Drug: Gadolinium

INTERVENTIONS:
Drug: Iodohippurate — An injection of non-radioactive iodohippurate (0.07 mL/kg) will be administered to determine renal plasma flow (RPF)
  Other Names: RPF filtration
  Groups: Sepsis with Severe AKI
Procedure: 24 hour ambulatory Blood Pressure — Ambulatory blood pressure (BP) monitoring will be performed using a commercially available device (TIBA Ambulo 2400) for 24 hours with measurements every 30 minutes while awake and every hour during sleep.
Procedure: Peripheral Arterial Tonometry — The peripheral arterial tonometry (PAT) device measures changes in the cutaneous circulation that correlate with flow-mediated dilatation.
Procedure: Pulse Wave Velocity — Carotid-femoral and carotid-radial pulse wave velocities (PWV), validated markers of individual cardiovascular risk, will be determined by applanation tonometry using SphygmoCorVx technology (AtCor Medical). PWV is an index of the overall stiffness of a vascular segment between measurement sites 59. Thus, while carotid-femoral PWV is an index of the overall stiffness of proximal (central) arteries, the overall stiffness of peripheral arteries contributes relatively more to carotid-radial PWV.
Drug: Gadolinium — Dotarem Gadolinium (GD)- Gadoterate Meglumine (0.07 to 0.14 mL/kg) will be used to determine GFR.
  Other Names: Dotarem Gadolinium (GD); Glomerular Function Rate (GFR) filtration

SUMMARY:
Sepsis is the most common cause of childhood death worldwide. Millions of children survive, but are left with impaired health. Sepsis-related Acute Kidney Injury (sAKI) is increasingly recognized as a significant factor associated with long-term mortality among different patient populations. Renal dysfunction and subsequent chronic kidney disease is implicated in the development of hypertension and cardiovascular disease. The investigators overall hypothesis is that, in the pediatric population, sepsis-related AKI will have unrecognized, long-term consequences with regard to kidney function, endothelial function, blood pressure control, and overall health.

DETAILED DESCRIPTION:
This will be a two-arm cross-sectional control-cohort outpatient evaluation. Subjects with sAKI and control subjects (age and gender matched) will be recruited from neurology service. Subjects will be asked to come in to the Clinical Research Center for 24-hour monitoring and participate in the outpatient study where urinary and serum studies to measure glomerular filtration rate, renal plasma flow followed by blood pressure monitoring, peripheral arterial and applanation tonometry.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Ability to assent (age 7-17 at time of participation in the study)
* If taking antihypertensive medication, prescribing practitioner's written approval to participate

For sAKI patients:

* Hospitalization with a diagnosis of sepsis from 1998-2014
* Severe AKI as defined by the pEDRIFLE criteria during incident sepsis admission
* Participation in cognitive survey study with completion of the PedsQL survey

For healthy control patients:

• Patients from the neurology service undergoing MRI with gadolinium as a part of their clinical care

Exclusion Criteria:

For all patients:

* Known pre-existing CKD as defined by history of kidney transplant or long-term dialysis
* Age greater than 17 years at the time of incident sepsis admission
* AKI from primary kidney disease including acute glomerulonephritis and obstructive uropathy
* Pregnancy at the time of enrollment
* Known or suspected allergy to gadolinium based contrast
* Known or suspected allergy to iodohippurate will be excluded from RPF measurement with iodohippurate
* Heart failure or condition whereby the administration of 0.9% normal saline would be contraindicated
* If taking antihypertensive medication, lack of prescribing practitioner's written approval to participate

For healthy control patients:

* Chronic kidney disease
* History of acute kidney injury or GFR <100 History of chronic illnesses deemed to predispose to renal or cardiovascular dysfunction or abnormalities Suspicion of infection
* Neuro-vascular history such as encephalitis, meningitis, vascular anomalies of the brain or spinal cord or cerebrovascular infarct or ischemia will be excluded .
* No indication for gadolinium administration for MRI

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Contact and enroll subjects with severe sepsis related AKI subjects without sepsis related AKI and a sample of age and sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Glomerular Function Rate (GFR) filtration | Day 2
  Magnevist Gadolinium (GD)-diethylene-triamine-pentaacetic acid-bis-oleate (0.07 to 0.14 mL/kg) will be used to determine GFR.
Renal plasma flow (RPF) filtration | Day 2
  An injection of non-radioactive iodohippurate (0.07 mL/kg) will be administered to determine renal plasma flow (RPF) filtration.
Proteinuria will be measured in the urine | Day 2
  Proteinuria may be a sign of renal (kidney) damage. Since serum proteins are readily reabsorbed from urine, the presence of excess protein indicates either an insufficiency of absorption or impaired filtration. People with diabetes may have damaged nephrons and develop proteinuria.
Cystatin C will be measured in the blood | Day 2
  Cystatin C can be measured in a random sample of serum (the fluid in blood from which the red blood cells and clotting factors have been removed) using immunoassays such as nephelometry or particle-enhanced turbidimetry.

SECONDARY OUTCOMES:
24 hour ambulatory Blood Pressure | 24 hours
  Ambulatory blood pressure (BP) monitoring will be performed using a commercially available device (TIBA Ambulo 2400) for 24 hours with measurements every 30 minutes while awake and every hour during sleep.
Peripheral Arterial Tonometry | 24 hours
  The peripheral arterial tonometry (PAT) device measures changes in the cutaneous circulation that correlate with flow-mediated dilatation.
Pulse wave velocity | 24 hours
  Carotid-femoral and carotid-radial pulse wave velocities (PWV), validated markers of individual cardiovascular risk, will be determined by applanation tonometry using SphygmoCorVx technology (AtCor Medical). PWV is an index of the overall stiffness of a vascular segment between measurement sites 59. Thus, while carotid-femoral PWV is an index of the overall stiffness of proximal (central) arteries, the overall stiffness of peripheral arteries contributes relatively more to carotid-radial PWV.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Carmelle Elie, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States